CLINICAL TRIAL: NCT03541941
Title: Exparel vs. Bupivacaine Hydrochloride vs. Placebo for Transversus Abdominis Plane Blocks During Open Retromuscular Hernia Repair
Brief Title: Exparel vs. Bupivacaine Hydrochloride vs. Placebo for Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Michael Rosen, Staff Surgeon, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-133
Record Dates: First submitted 2018-05-04; First posted 2018-05-31 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Analgesia, Postoperative
Keywords: Liposomal Bupivacaine; Exparel; Transversus Abdominis Plane block; Hernia
MeSH Terms: conditions — Agnosia; Hernia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exparel (Experimental): Solution of 266mg of Exparel + 150mg Bupivacaine HCL + 40cc normal saline= 120cc administered through a transversus abdominis plane block performed intraoperatively by the surgeon under direct visualization
  Interventions: Drug: Exparel; Drug: Bupivacaine Hcl 0.25% Inj
- Bupivacaine Hcl 0.25% Inj (Active Comparator): Solution of 150mg Bupivacaine HCL expanded with 60cc of normal saline=120cc administered through a transversus abdominis plane block performed intraoperatively by the surgeon under direct visualization
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj
- Placebo (Placebo Comparator): 120 cc of normal saline administered through a transversus abdominis plane block performed intraoperatively by the surgeon under direct visualization
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exparel — Solution of: 266mg of Bupivacaine Liposome Injectable Suspension (Exparel) mixed with 150mg of Bupivacaine Hydrochloride 0.25% expanded with 60cc of Normal Saline (Nacl0.9%) administered intraoperatively through a transversus abdominis plane (TAP) block
  Arms: Exparel
Drug: Bupivacaine Hcl 0.25% Inj — Solution of: 150mg of Bupivacaine Hydrochloride 0.25% expanded with 60cc of Normal Saline (Nacl0.9%) administered intraoperatively through a transversus abdominis plane (TAP) block
  Arms: Bupivacaine Hcl 0.25% Inj; Exparel
Drug: Placebo — Normal saline administered intraoperatively through a transversus abdominis plane (TAP) block
  Arms: Placebo

SUMMARY:
Patients usually experience some level of pain after their hernia repair. To control pain after the operation, surgeons have many options. One of them is to make some injections of pain blocker medications into the nerves that are responsible for the sensations the abdominal wall.This procedure is called TAP block (transversus abdominis place block). These medications are called local anesthetics, and there is a variety of medications that can be used. One of such medications is called Exparel® (Liposomal Bupivacaine). Exparel® has the potential benefit of lasting more hours than regular anesthetics. Although this drug is being used with increasing frequency, the investigators do not have good quality studies investigating the benefits of using this medication during a hernia repair, especially when compared to other types of local anesthetics (Bupivacaine Hydrochloride) or when compared to not injecting this medication at all. This study aim to investigate if Exparel®, when injected in the nerves of the abdominal wall during hernia repair can: (1) reduce the dose of additional opioid medications (morphine and similar) needed to achieve good pain control and (2) result in lower pain scores. The hypothesis is that Exparel® will result in a 30% decrease in the total requirements for opioid medications during the first 72 hours after surgery. Patients will be randomized to receive either Exparel®+Bupivacaine Hydrochloride, Bupivacaine Hydrochloride or Placebo (normal saline) during the operation through a TAP block. All patients will receive a patient controlled analgesia device after the operation, where patients can simply push a button every time they feel pain and the device will administer a dose of opioid medications. The investigators of the study will record the necessary amount of opioids used by the patients to achieve good pain control and also record pain scores several times during hospital stay.

DETAILED DESCRIPTION:
This will be a double-blind, 3-arm, randomized controlled trial with a treatment 1: treatment 2: control allocation ratio of 1:1:1. Primary outcomes of interest are opioid requirements and pain scores over initial 72 hours of the postoperative period. Opioid requirements will be assessed by measuring the cumulative dose of opioids administered intravenously (infused through a patient-controlled analgesia device as well as the quantity of opioids administered intravenously as rescue, if needed) and the quantity of opioids administered through oral preparations. This will be assessed at time points: while patients are at the post-anesthesia care unit (PACU), at postoperative days 1(24h±4 hours), 2(48h±4 hours), 3(72h±4 hours) and at the date of hospital discharge. The total dose of opioids used at each time point will be recorded and converted into morphine equivalents for standardization and analysis. The cumulative dose of opioids from 0 hours to 72 hours after the operation and for the total hospital length of stay will be recorded. In addition, the dose of opioids administered intra-operatively by the anesthesiologist, time for first oral opioid dose over the first 72 hours (discontinuation of PCA), and the percentage of patients not requiring opioids over the first 72 hours will also be recorded.

Pain scores will be determined using a 100mm visual analog scale (VAS). The VAS is a 100mm horizontal line with two endpoints: 0 (no pain) and 100 (worst imaginable pain). Pain scores will be assessed at baseline during preoperative evaluation, at the PACU, at postoperative days 1(24h±4 hours), 2(48h±4 hours), 3(72h±4 hours), and at the time of hospital discharge.

Additional pain scores will be obtained using the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey at baseline and 30-day follow-up. This survey will be completed by patients in person during enrollment and 30-day follow-up. Secondary outcomes of interest include the length of hospital stay and Patient-Reported Quality of Life (PRQOL). Both information is already routinely collected through the Americas Hernia Society Quality Collaborative (AHSQC). Length of hospital stay will be recorded in days. PRQOL will be assessed using the Hernia-Related Quality-of-Life survey (HerQLes). The HerQLes is a 12-item, validated, hernia-specific survey that assesses quality of life through abdominal wall function after ventral hernia repair. HeQLes scores will be assessed at baseline and 30 days after the operation.

All patients will undergo the same operation, under a standard of care protocol. Skin preparation, hair removal, perioperative antibiotics and venous thromboembolism prophylaxis will be performed per Surgical Care Improvement Project protocol guidelines. The procedure will be performed through a midline incision. Upon entering the abdominal cavity, all adhesions between intra-abdominal contents and the anterior abdominal wall are routinely lysed using sharp dissection. When present, hernia contents are reduced back to the cavity. At the end of adhesiolysis, the surgeon will ask the OR nurse to contact the investigational pharmacy via telephone, who will randomize the subject. The investigational pharmacy will be responsible for preparing and dispensing the assigned intervention. The OR nurse will receive the drug from the investigational pharmacy in a standardized bag and will dispense it to the surgeon at the time of the TAP block. Neither the surgeon nor other members of the surgical team will be informed about which of the interventions were assigned to the specific patient. Electronic medical records will contain the information: "Patient was randomized and assigned to receive intervention according to randomization performed by investigational pharmacy." Retromuscular hernia repair is performed initially incising the posterior rectus sheath just lateral to the linea alba. The release will be performed at least 5 cm above and below the fascial defect, and retrorectus dissection is carried out laterally in the direction of the linea semilunaris. If deemed necessary, a posterior component separation will be performed by incising the posterior lamella of the internal oblique, dividing the fibers of the transversus abdominis muscle and dissecting the preperitoneal and retroperitoneal spaces of the lateral abdominal wall laterally.

At the end of the myofascial release, randomization will occur and the assigned intervention drug will be dispensed in syringes to the surgeon who will perform the perform a TAP block under direct visualization. Patients will be randomized using a computer-generated random allocation sequence, by the investigational pharmacy personnel.

Injections of the designated drug (group 1, 2 or 3) will be performed under direct visualization by the attending surgeon, in 5 vertical levels, to the thoracoabdominal nerves (from T7 to T11).

The interventions are:

* Treatment 1- Administration of a solution of Exparel® combined with Bupivacaine Hydrochloride 0.25% and normal saline, through a bilateral TAP block performed intraoperatively by the attending surgeon, during open ventral hernia repair;
* Treatment 2: Administration of a solution of Bupivacaine Hydrochloride 0.25% and normal saline, through a bilateral TAP block, performed intraoperatively by the attending surgeon, during open ventral hernia repair ;
* Control (Placebo): administration of normal saline through a bilateral TAP block performed intraoperatively by the attending surgeon, during open ventral hernia repair.

The posterior sheath will be reapproximated, and a standard piece of polypropylene mesh will be placed in the retromuscular space.

Mesh type will be defined by the surgeon intraoperatively according to the patient and hernia-specific variables. Mesh fixation will be performed circumferentially using mechanical sutures. Closed suction drains will be placed above the mesh and in the subcutaneous space, and the timing of removal will be based on the surgeon's standard practice. Fascial closure and management of wound dressings will also follow the surgeon's standard practice.

For postoperative analgesia, all patients will also receive a patient-controlled analgesia (PCA) device according to the standard of care; preferably:

• Hydromorphone HCL 0.5mg/ml (Dilaudid®, Purdue Pharmaceuticals, Stamford, CT) in 100ml of normal saline, with no basal rate infusion, a patient bolus dose of 0.2-0.4mg, bolus interval of 6 minutes (maximum 10 doses per hour).

To ensure the comfort and adequate pain postoperative pain control, additional intravenous or oral opioids are allowed in the protocol, to be administered for breakthrough pain (as needed). Subjects should only receive rescue medication upon request, and for pain control.

Estimated patient accrual time is 2 years with data collection to occur over 30 days from randomization of each patient. Data analysis and manuscript production will occur within 6 months of the completion of data collection.

As with any surgical procedure, patients may experience pain, bleeding, and discomfort. Common occurrences following hernia repair include seroma, hematoma, inflammation, wound dehiscence, and infection. Risks of Bupivacaine Hydrochloride include allergic reactions, arrhythmias, chest pain or pressure, dizziness, confusion, restlessness, tinnitus, blurred vision, dyspnea, seizures, nausea, emesis, and lethargy. Risks of Exparel® include nausea, vomiting, constipation, as well as (rarely) seizures and cardiac arrest. Patients receiving placebo intraoperatively will not necessarily experience higher levels of pain, as all individuals, regardless of intervention arm, will be provided a multimodal pain management regimen with patient-controlled analgesia postoperatively. There are no direct benefits to subjects for participation in this study. Subject participation will, however, help physicians and hospital administrators better understand the outcomes of Exparel® use concerning postoperative pain management and its influence on opioid consumption, hospital length of stay and quality of life. Patients are under no obligation to participate in this study. A member of the research team will discuss all available surgical options with patients. It will be emphasized that refusal to participate in this study will not impact any patient's ability to receive surgical care. There will be no payment for the subjects for the participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Primary Ventral or Incisional Hernias
* Scheduled to undergo hernia repair through an open approach
* Hernia repair performed in an elective setting
* Hernia repair performed through a midline incision
* Hernia repair performed in a clean wound
* Hernia repair performed with mesh placed in the retromuscular position

Exclusion Criteria:

* patients with less than 18 years old of age
* patients scheduled to undergo a minimally invasive hernia repair
* patients where hernia repair is planned to be performed with mesh placement in a different position than retromuscular
* patient undergoing hernia repair with a clean-contaminated, contaminated or infected wound
* patients undergoing hernia repair in an non-elective fashion
* patients with allergy, hypersensitivity or contraindication to bupivacaine
* patients with history of chronic liver disease with moderate or severe impairment in liver function defined as a Child-Pugh class B or C
* patients with chronic kidney disease on dialysis
* chronic opioid users, defined as daily or near daily use of opioids for at least 90 days in the past year
* patients unable to provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Rosen, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Comprehensive Hernia Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fafaj A, Krpata DM, Petro CC, Prabhu AS, Rosenblatt S, Tastaldi L, Alkhatib H, Tu C, Zolin SJ, Thomas JD, Costanzo AM, Rosen MJ. The Efficacy of Liposomal Bupivacaine on Postoperative Pain Following Abdominal Wall Reconstruction: A Randomized, Double-blind, Placebo-controlled Trial. Ann Surg. 2022 Aug 1;276(2):224-232. doi: 10.1097/SLA.0000000000004424. Epub 2020 Dec 2. PMID 33273351

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Started | 57 | 55 | 52
Completed | 57 | 55 | 52
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo | Total
Number analyzed (Participants) | 57 | 55 | 52 | 164
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.0 [52.0 to 68.0] | 58.0 [53.0 to 69.0] | 60.0 [54.0 to 65.0] | 59.0 [53.0 to 67.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 29 | 81
  Male | 32 | 28 | 23 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 57 | 55 | 52 | 164

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Opioid Requirements for 72 Hours After Surgery
Description: Measured in milligrams or micrograms as appropriate and converted to oral morphine equivalent daily dose. The cumulative dose of opioids administered intravenously (infused through a patient-controlled analgesia device as well as the quantity of opioids administered intravenously as rescue, if needed) and the quantity of opioids administered through oral preparations will be recorded. Such assessment will be performed at the 3rd postoperative day (72 hours of operation).
Time Frame: Measured from end of surgery until 72 hours after the surgery
Measure: Mean (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
mg morphine equivalents/day | 325 (225) | 350 (284) | 310 (272)

2. Primary Outcome: Cumulative Opioid Requirements at Postoperative Day 0
Description: Measured in milligrams or micrograms as appropriate and converted to oral morphine equivalent daily dose. The cumulative dose of opioids administered intravenously (infused through a patient-controlled analgesia device as well as the quantity of opioids administered intravenously as rescue, if needed) and the quantity of opioids administered through oral preparation will be measured at postoperative day 0 (day of surgery).
Time Frame: From end of surgery until the end of postoperative day 0 (23:59pm of postoperative day 0)
Measure: Mean (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
mg morphine equivalents/day | 68.3 (49.8) | 77.1 (62.5) | 74.5 (54)

3. Primary Outcome: Cumulative Opioid Requirements at Postoperative Day 1
Description: Measured in milligrams or micrograms as appropriate and converted to oral morphine equivalent daily dose. Cumulative dose of opioids administered intravenously (infused through a patient-controlled analgesia device as well as the quantity of opioids administered intravenously as rescue, if needed) and the quantity of opioids administered through oral preparations, measured at postoperative day 1
Time Frame: From 00:00am of postoperative day 1 until (23:59pm of postoperative day 1)
Measure: Mean (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
mg morphine equivalents/day | 116 (81.7) | 116 (100) | 105 (92.1)

4. Primary Outcome: Cumulative Opioid Requirements at Postoperative Day 2
Description: Measured in milligrams or micrograms as appropriate and converted to oral morphine equivalent daily dose. Cumulative dose of opioids administered intravenously (infused through a patient-controlled analgesia device as well as the quantity of opioids administered intravenously as rescue, if needed) and the quantity of opioids administered through oral preparations, measured at postoperative day 2
Time Frame: From 00:00 of postoperative day 2 until 23:59pm of postoperative day 2
Measure: Mean (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
mg morphine equivalents/day | 79.9 (69.8) | 96.7 (94) | 79.9 (97.4)

5. Primary Outcome: Cumulative Opioid Requirements at Postoperative Day 3
Description: Measured in milligrams or micrograms as appropriate and converted to oral morphine equivalent daily dose. Cumulative dose of opioids administered intravenously (infused through a patient-controlled analgesia device as well as the quantity of opioids administered intravenously as rescue, if needed) and the quantity of opioids administered through oral preparations, measured at postoperative day 3
Time Frame: From 00:00 of postoperative day 3 until 23:59pm of postoperative day 3
Measure: Mean (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
mg morphine equivalents/day | 60.9 (56.4) | 60.4 (68.5) | 50.9 (68.9)

6. Secondary Outcome: Opioid Requirements for Total Length of Hospital Stay
Description: Cumulative dose of opioids administered intravenously (infused through a patient-controlled analgesia device as well as the quantity of opioids administered intravenously as rescue, if needed) and the quantity of opioids administered through oral preparations administered during the entire length of hospital stay. Measured in milligrams or micrograms as appropriate and converted to oral morphine equivalent daily dose.
Time Frame: Measured from end of surgery until the time of hospital discharge, up to a maximum of 6 days
Measure: Mean (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
mg morphine equivalents/day | 50.5 (17.2) | 50.1 (19.1) | 51.0 (20.5)

7. Secondary Outcome: Pain Scores at Postoperative Day 0
Description: Measured using a 100mm Visual Analog Scale, at the end of the first of postoperative day 0 (day of surgery).
  The scale ranges from 0mm (No pain) to 100mm (Pain as bad as it could possibly be). A paper-based version of the VAS will be used, containing a 100mm line, where the left-end (0mm) contains the sentence "No Pain" and in the right-end (100mm) contains the sentence "Pain as bad as it could possibly be". Patients will be asked to indicate on the line where the pain is in relation to the two extremes. This will be performed with a pen. Measure with a ruler will be performed from the left hand side to the mark and this will be recorded in mm. Lower values represent less pain and higher values represent more pain. There are no subscale components for this measurement.
Time Frame: Measured once, from end of surgery until the end of postoperative day 0 (23:59pm of the day of surgery)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
score on a scale | 20.0 [1.00 to 57.0] | 16.0 [2.00 to 42.5] | 21.5 [2.00 to 32.2]

8. Secondary Outcome: Pain Scores at Postoperative Day 1
Description: Measured using a 100mm Visual Analog Scale, at the end of the postoperative day 1.
  The scale ranges from 0mm (No pain) to 100mm (Pain as bad as it could possibly be). A paper-based version of the VAS will be used, containing a 100mm line, where the left-end (0mm) contains the sentence "No Pain" and in the right-end (100mm) contains the sentence "Pain as bad as it could possibly be". Patients will be asked to indicate on the line where the pain is in relation to the two extremes. This will be performed with a pen. Measure with a ruler will be performed from the left hand side to the mark and this will be recorded in mm. Lower values represent less pain and higher values represent more pain. There are no subscale components for this measurement.
Time Frame: Measured once, from 00:00am of postoperative day 1 until the end of postoperative day 1 (23:59pm of postoperative day 1)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
score on a scale | 58.0 [27.0 to 73.0] | 49.0 [32.5 to 70.5] | 42.5 [23.0 to 60.0]

9. Secondary Outcome: Pain Scores at Postoperative Day 2
Description: Measured using a 100mm Visual Analog Scale, at the end of the postoperative day 2 The scale ranges from 0mm (No pain) to 100mm (Pain as bad as it could possibly be). A paper-based version of the VAS will be used, containing a 100mm line, where the left-end (0mm) contains the sentence "No Pain" and in the right-end (100mm) contains the sentence "Pain as bad as it could possibly be". Patients will be asked to indicate on the line where the pain is in relation to the two extremes. This will be performed with a pen. Measure with a ruler will be performed from the left hand side to the mark and this will be recorded in mm. Lower values represent less pain and higher values represent more pain. There are no subscale components for this measurement.
Time Frame: Measured once, from 00:00am of postoperative day 2 until the end of postoperative day 2 (23:59pm of postoperative day 2)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
score on a scale | 56.0 [32.0 to 69.0] | 39.0 [25.5 to 56.5] | 42.5 [21.5 to 56.2]

10. Secondary Outcome: Pain Scores at Postoperative Day 3
Description: Measured using a 100mm Visual Analog Scale, at the end of the postoperative day 3 The scale ranges from 0mm (No pain) to 100mm (Pain as bad as it could possibly be). A paper-based version of the VAS will be used, containing a 100mm line, where the left-end (0mm) contains the sentence "No Pain" and in the right-end (100mm) contains the sentence "Pain as bad as it could possibly be". Patients will be asked to indicate on the line where the pain is in relation to the two extremes. This will be performed with a pen. Measure with a ruler will be performed from the left hand side to the mark and this will be recorded in mm. Lower values represent less pain and higher values represent more pain. There are no subscale components for this measurement.
Time Frame: Measured once, from 00:00am of postoperative day 3 until the end of postoperative day 3 (23:59pm of postoperative day 3)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
score on a scale | 46.0 [26.0 to 74.0] | 45.0 [24.0 to 60.0] | 40.0 [22.0 to 51.5]

11. Secondary Outcome: Length of Hospital Stay
Description: Measured in days, being the difference from day of surgery until the day of hospital discharge.
  The scale ranges from 0mm (No pain) to 100mm (Pain as bad as it could possibly be). A paper-based version of the VAS will be used, containing a 100mm line, where the left-end (0mm) contains the sentence "No Pain" and in the right-end (100mm) contains the sentence "Pain as bad as it could possibly be". Patients will be asked to indicate on the line where the pain is in relation to the two extremes. This will be performed with a pen. Measure with a ruler will be performed from the left hand side to the mark and this will be recorded in mm. Lower values represent less pain and higher values represent more pain. There are no subscale components for this measurement.
Time Frame: From the day of surgery until the day of hospital discharge, up to a maximum of 30 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
Days | 5.00 [5.00 to 7.00] | 5.00 [5.00 to 6.00] | 5.00 [4.00 to 6.00]

12. Secondary Outcome: 30-day Pain Scores
Description: Measured using the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey. This survey has 3 questions:(1) How intense was your pain as its worst? (2) How intense was your average pain? and (3) What is your level of pain right now?. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score, sum of the values for each question is performed; lowest possible raw score is 3 and highest possible raw score is 15.A raw score of 10 converts to a T-score of 54.5 with a standard error (SE) of 2.9. Thus, the 95% confidence interval around the observed score ranges from 48.8 to 54.5 (T-score + (1.96*SE) or 54.5 + (1.96*2.9). A score of 50 is the average for the United States general population with a standard deviation of 10. For negatively-worded concepts like Pain Intensity, a T-score of 60 is one SD worse than average. By comparison, a Pain Intensity Tscore of 40 is one SD better than average.
Time Frame: Measured during the 30-day follow-up visit, expected to occur 30-days after the day of surgery, up to a maximum of 90 days
Measure: Median (Inter-Quartile Range); unit: T-Score
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
T-Score | 19.0 [4.00 to 50.0] | 16.5 [4.00 to 50.0] | 11.0 [3.00 to 26.0]

13. Secondary Outcome: 30-day Patient-Reported Quality of Life
Description: Measured using the Hernia Related Quality of Life survey (HerQLes) during the 30-day follow-up visit. The HerQLes is a valid and reliable hernia-specific quality of life measure. Each questions has 6 response options ranging in value from one to six. To find the raw score for the HerQles, a sum of the values of the response to each question is performed. For example, the lowest possible score is 12; the highest possible score is 72. All questions must be answered to provide a valid score. Mean and standard deviations of the scores of the entire study population will be calculated. Next, the Z score will be calculated as follows:
  (Raw score-mean) / Standard Deviation. Next step is to calculate the Standard Score, as follows: (-(Z score)*Mean)+Standard Deviation. The standard score will be used for comparisons and reports, and should provide a value ranging from 0 to 100. Lower scores means lower quality of life and higher scores means higher quality of life.
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
Number analyzed (Participants) | 57 | 55 | 52
Z-Score | 46.9 (29.1) | 38.4 (24.3) | 45.2 (23.5)

ADVERSE EVENTS:
Time Frame: 30 days following surgery
Arm/Group | Exparel | Bupivacaine Hcl 0.25% Inj | Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/55 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/57 | 2/55 | 0/52
Other Adverse Events (participants affected / at risk) | 15/57 | 17/55 | 7/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel (N=57) | Bupivacaine Hcl 0.25% Inj (N=55) | Placebo (N=52)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel (N=57) | Bupivacaine Hcl 0.25% Inj (N=55) | Placebo (N=52)
Ileus (Gastrointestinal disorders) | 14 (14) | 11 (11) | 6 (6)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03541941/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03541941/ICF_001.pdf